CLINICAL TRIAL: NCT01728272
Title: Influence of CPB and Mini CPB to the Absorption of the Metoprolol After CABG
Brief Title: Influence of CPB and Mini CPB to the Absorption of the Metoprolol
Acronym: Minimeto
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5101066
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Drug Absorption
Keywords: metoprolol, atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- blood concentration of metoprolol (Experimental): how does off-pump miniperfusion and perfusion CABG influence the absorption of metoprolol after CABG
  Interventions: Drug: blood concentration of metoprolol

INTERVENTIONS:
Drug: blood concentration of metoprolol — measure blood concentration of metoprolol

SUMMARY:
Influence of perfusion, miniperfusion and off pump coronary artery bypass grafting to the absorbtion of metoprolol postoperatively, hypothesis in that miniperfusion and off pump surgery does not decrease absorbtion of the metoprolol compared to conventional pefusion.

DETAILED DESCRIPTION:
Influence of perfusion, miniperfusion and off pump coronary artery bypass grafting to the absorbtion of metoprolol postoperatively, hypothesis in that miniperfusion and off pump surgery does not decrease absorbtion of the metoprolol compared to conventional pefusion.

Blood samples for concentration of metoprolol are taken preoperaively, 1. and 3. day after operation, before and 10 times after intake of 50 mg metoprolol.

Sudy is randomized into 3 groups: 1. Miniperfusion n.15 2. Perfusion n.15 3. offpump n.15

ELIGIBILITY:
Inclusion Criteria: elective CABG patient -

Exclusion Criteria: contraindication to metoprolol

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
absorbtion of the metoprolol | one year
  absorbtion of the metoprolol, blood samples are taken centrifuged, frozed and analyzed

SECONDARY OUTCOMES:
atrial fibrillation | one year
  is there correlation of incidence of the postopeative AF and absorbtion of the metoprolol

OTHER OUTCOMES:
recovery from rocedure | one year
  How does gereral recovery correlate between randomized groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Kuopio, Finland